CLINICAL TRIAL: NCT07127107
Title: Effect of Manual Therapy on Migraine in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Mohamed Yassen, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005876
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-steroidal anti-inflammatory drugs (NSAIDs) group (Active Comparator): The participants will receive non-steroidal anti-inflammatory drugs (NSAIDs) to relieve the pain and symptoms of a migraine attack and help prevent further migraine attacks
  Interventions: Drug: Non-steroidal anti-inflammatory drugs (NSAIDs)
- Manual therapy group and non-steroidal anti-inflammatory drugs (NSAIDs) group (Experimental): The participants will receive the same medical treatment (non-steroidal anti-inflammatory drugs (NSAIDs)) plus manual therapy techniques for 3 times per week for 8 weeks.
  Interventions: Drug: Non-steroidal anti-inflammatory drugs (NSAIDs); Other: Manual therapy techniques

INTERVENTIONS:
Drug: Non-steroidal anti-inflammatory drugs (NSAIDs) — For mild and moderate migraines e.g Ibuprofen and aspirin.
  * Aspirin: Peroral (PO) tablet with standard dosages of 325 mg, 500 mg, and 400 mg effervescent; treatment dosage of up to 1000 mg
  * Ibuprofen: PO tablet with standard dosages of 200 mg, 400 mg, 600 mg, and 800 mg; treatment dosage of 200 to 800 mg
Other: Manual therapy techniques — Cranial manipulative osteopathy: Tension release of cranial sutures is applied while the patient in supine lying position, a pressure of 200g to3kg is applied with both thumbs for 30-40 sec or till release occurs. it includes:
  1. Coronal suture The head is directed to one side and the pressure is applied with both thumbs directed parallel to each otheralong the coronal suture.
  2. Sagital suture distraction The head is in the central position and the pressure is applied with both thumbs directed parallel to each other along the sagittal suture.
  3. Squamous suture distraction The head is directed to one side and the pressure is applied with both thumbs parallel along the squamous suture.
  4. Lamboidal suture distraction:
     The head is directed to one side and the thumbs directed parallel to each other along the lamboidal suture.
  5. Occipitomastoid suture distraction The head is directed to one side and both thumbs directed parallel to each other along occipitomastoid suture.
  Arms: Manual therapy group and non-steroidal anti-inflammatory drugs (NSAIDs) group

SUMMARY:
The purpose of the study is to determine the effect of manual therapy on migraine in postmenopausal women.

DETAILED DESCRIPTION:
Menopause is a period of great changes to women's bodies and minds. Alterations to body image and emotions, psychological adjustment to a new phase of life and worries about the higher prevalence of severe diseases and cognitive dysfunction all contribute towards negatively affecting the quality of life of menopausal patients. Symptoms that are typical of hormonal deprivation and aging are prevalent and distressful to many, often requiring individual counseling and specific therapies. Some of the symptoms are manageable and headache is certainly a modifiable parameter if given the appropriate treatment. About one third of the women had experienced worsening of their primary headaches after their last menstrual period, which contradicts the popular belief that "after menopause the headache gets better.

Migraine is a severe headache often felt as a throbbing pain - and usually occurring on one side of the head. It often comes with nausea or vomiting, and a heightened sensitivity to light or sound. The headache is such that it stops doing what is normally do and can last from four to 72 hours .

Soft tissue massage of the paraspinal muscles, jaw muscles will all help decrease the muscle spasm of tension headaches. Joint Manipulation: this can be done with manipulative techniques or gentle articulation techniques to encourage joint release and movement By manipulating the bones of skull and the dura mater that is a membrane just below the skull, craniosacral therapy also relieves arterial pressure to ease pain.

There is dearth of knowledge regarding the effect of manual therapy on migraine in postmenopausal women. This study, therefore, contributes valuable insights to a relatively unexplored area of

ELIGIBILITY:
Inclusion Criteria:

* All women are postmenopausal at least one year following last menstruation.
* They are suffering from migraine.
* Their ages will range from 50 to 60 years old.
* Their body mass index (BMI) will not exceed 30 Kg/m2.
* Women with regular or irregular attacks of migraine.

Exclusion Criteria:

* Artificial or premature menopause
* Recent head trauma.
* Cerebral aneurysm or rupture.
* Tumors.
* Acute intracerebral bleeding.
* Hormonal replacement therapy.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | 8 weeks
  Pressure algometry (PA) is a method described to objectify pressure pain threshold PPT.
  Application:
  * Frontal muscle (2 cm above the surfacing of the supra orbital branch of the trigeminal nerve) Medium temporalis muscle (located 2 cm to the lateral rim of the eyebrow)
  * Masseter muscle (origin: anterior rim of the surface portion of the muscle; insertion: lower most prominent region identified by manual palpation during maximal dental clenching, and belly: the mid-point between the origin and the insertion) ;
  * Trapezius (insertion: the point immediately below the occipital bone, located in the sub-occipital region; upper fibers: mid-point between the spinous process of seventh cervical vertebrae (C 7) and the acromion);
  * Sternocleidomastoid muscle (upper portion: fibers below the mastoid process)
  * PPT levels were obtained in three consecutive series bilaterally
Migraine disability assessment Questionnaire : | 8 weeks
  Migraine Disability Assessment (MIDAS) questionnaire was designed to be brief, self-administered, and easy to score. It assesses not only missed days of activity, but also days in which productivity is reduced by at least half.
  The MIDAS score is derived as the sum of missed days and days when productivity was reduced by at least half for work outside the home and household work, as well as missed days of nonwork activities (family, social, and leisure) during a 3-month period. The score, therefore, has units of lost days. Physicians graded each patient for pain level (mild, moderate, or severe), level of disability (none, mild, moderate, or severe), and need for medical care (from 0 [lowest] to 100 [highest]).
The blink reflexometer | 8 weeks
  It is an electrodiagnostic test that evokes the corneal reflex. It evaluates the integrity of the trigeminal and facial nerve. The supraorbital branch of the ophthalmic division of the trigeminal nerve constitutes the afferent arm, while the motor fibers of the facial nerve form the efferent arm of this reflex.Normally, as with the corneal reflex, the ipsilateral electrical stimulation of the trigeminal nerve will produce an eye blink bilaterally.
  The subject is supine and asked to stay relaxed with their eyes open or gently closed. The active electrode (A) is placed over the inferior aspect of the orbicularis oculus while the reference electrode (R) is placed either over the bony prominence of the zygomatic arch or the nose. The ground electrode (G) can be placed over the forehead or under the chin. Using a prong stimulator, each supraorbital nerve is stimulated and the response from the orbicularis oculus is recorded bilaterally.

SECONDARY OUTCOMES:
Migraine-Specific Quality of Life Questionnaire (MSQv2.1) | 8 weeks
  The MSQv2.1 measures quality of life among migraine patients during the past 4 weeks. It has three scales:(1) Role Restrictive (RR, original named Role Function-Restrictive in MSQv1), which includes seven items that assess how patients' performance of normal activities is limited by migraine; (2) Role Preventive (RP, original named Role Function-Preventive), which consists of four items that assess how patients' performance of normal activities is interrupted by migraines; and (3) Emotion Function (EF), which consists of three items that assess the impact of migraine on the respondent's emotions (e.g., frustration or helplessness). The item responses range from one to six (1 = "None of the time;" 2 = "A little bit of time;" 3 = "Some of the time;" 4 = "A good bit of the time;" 5 = "Most of the time;" 6 = "All of the time"). All items are reverse-coded, and standardized to a 0-100 scale. Thus, higher scale scores indicate better migraine-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mahmoud, Professor, Study Director — Cairo University; Amel Youssef, Professor, Study Chair — Cairo University
Locations (1):
- Marwa Mohamed Mohamed Yassen, Cairo, Egypt